CLINICAL TRIAL: NCT01443247
Title: Role of Andi-d in Dengue Fever: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Deepak Thakur, junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dengue fever pgimer trial
Record Dates: First submitted 2011-09-25; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — RHO(D) antibody; gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- platelet support + anti-d (Experimental)
  Interventions: Drug: anti-d
- platelet support (No Intervention)
  Interventions: Drug: anti-d

INTERVENTIONS:
Drug: anti-d — intervention group received injection anti-d in dose of 50 µg/kg (250IU/kg) along with platelet concentrate while control ( non intervention ) group received platelet support only
  Other Names: winrho SDF

SUMMARY:
The purpose of this study is evaluate the role of anti-d in dengue fever.

DETAILED DESCRIPTION:
This study was conducted in pgimer. Patients presenting with fever and thrombocytopenia in emergency medical opd / medicine opd were screened and all dengue serology positive patients were evaluated for enrolment into the study. We had proposed to enroll 30 patients with diagnosed dengue haemorrhagic fever. the diagnosis of the dengue fever was based upon the clinical history ,general physical examination and the lab tests : thrombocytopenia ( platelet count ≤ 20,000 ) ,and a positive dengue serology.

STUDY DESIGN : It was an open label inteventional study . one group of 15 patients ( intervention group ) received platelet support along with injection anti-d in a dose of 50 µg/kg (250IU/kg) intravenously while the other group of 15 ( control group) received platelet support only . a base line platelet count of all the participant of both the study groups was taken and then the level of platelets at 12 , 24 , 36 , and 48hr post treatment initiation was noted. The patients were followed till the time of discharge .

ELIGIBILITY:
inclusion criteria:

* fever and thrombocytopenia with/without bleeding manifestations
* dengue serology positive patients
* platelet count ≤ 20,000/mm3
* Rh positive patients
* willing to give written informed consent

exclusion criteria:

* dengue serology positive but platelet count > 20,000/mm3
* Rh negative patients
* pregnant females

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
to see for the number of patients attaining a platelet count ≥ 50,000 /mm3 after 48 hours of administration of anti-d in the intervention arm | 1 YEAR

SECONDARY OUTCOMES:
the difference in two study arms with respect to: total volume of platelet concentrate transfused , duration of hospital stay , & severity of haemorrhagic manifestations | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: deepak thakur, md, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research , Chandigarh , India, Chandigarh, Chandigarh, India